CLINICAL TRIAL: NCT05233670
Title: Percutaneous Treatment of Iatrogenic False Femoral Aneurysms by Ultrasound-guided Thrombin Injection
Acronym: EGTI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EGTI
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Femoral; Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the 2000s, endovascular procedures have been expanding rapidly in multiple disciplines: cardiology, radiology, interventional neuroradiology, and of course vascular surgery. Most procedures are performed by puncture of the common femoral artery with introducers ranging in size from 4F to 26F for aortic procedures.

The most frequent complications of percutaneous punctures are false femoral aneurysms due to failure to close the arterial gap (up to 8% in some studies). A false aneurysm is a pocket of blood communicating with an artery and secondary to the rupture of the arterial wall. The blood is then contained by the adjacent structures and often a fibrous shell which distinguishes it from an aneurysm which retains the integrity of its wall.

The management of false femoral aneurysms is variable. Below 2 cm, monitoring may be performed with or without manual or ultrasound-guided compression. In case of persistence of the false aneurysm and/or complication, open surgery can be performed.

Endovascular treatment of false aneurysms was first proposed in 1986. Different endovascular techniques can be proposed to occlude false aneurysms such as the use of coils, biological glue, the use of arterial closure systems...

Echoguided injection of thrombin to occlude the false aneurysm in a manner has been published since the late 1990s. The treatment is evaluated as reliable and safe. A recent article in the EJVES (6) investigates the value of low-dose thrombin for this indication, and the results appear to be very encouraging for low-dose thrombin in false femoral aneurysms.

Thrombin injection for the treatment of iatrogenic false femoral aneurysms is the technique currently favoured by the vascular surgery team at the Paris Saint Joseph Hospital Group (GHPSJ). Open surgery is a second-line treatment and remains indicated in case of acute symptoms (radiculalgia, motor/sensory deficits; ischemia, skin necrosis), a false aneurysm that is too deep or without a neck, an infectious origin or a patient treated with dabigatran. Patients will be reviewed at 1 and 12 months according to the usual follow-up.

In this work, investigators will study the efficacy of false aneurysm closure using human thrombin injection. This work is intended to confirm previous work. A socio-economic study may be conducted in parallel. Follow-up after the use of percutaneous closure systems and in the context of bypass surgery may also be of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with iatrogenic false femoral arterial aneurysm, post arterial or venous puncture, following management for a diagnostic or therapeutic examination.
* Circulating false aneurysm confirmed by an imaging examination (echo-Doppler, angioscanner; angio-MRI).
* Indication for exclusion of false aneurysm
* False aneurysm treated at GHPSJ between 01/09/2020 and 31/12/2022 by thrombin injection

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients were or are referred for a post puncture false femoral aneurysm between 01/09/2020 and 31/12/2022.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy at 1 month of thrombin injection | Month 1
  This outcome corresponds to the percentage of false aneurysm thrombosis at 1 month.

SECONDARY OUTCOMES:
Intraoperative effectiveness of thrombin injection | Year 1
  This outcome corresponds to the number of intraoperative false aneurysm thrombosis and the number of false aneurysm thrombosis at 12 months.
Re-intervention | Year 1
  This outcome corresponds to the number of no re-intervention at the target lesion at 1 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yann GOUEFFIC, MD, PhD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Boge G, Laroche JP, Alric P. [Treatment of post-catheterization pseudoaneurysms by ultrasound-guided thrombin injection: A single-center experience and practical guideline]. J Med Vasc. 2017 Jul;42(4):198-203. doi: 10.1016/j.jdmv.2017.05.003. Epub 2017 Jun 28. French. PMID 28705337
- [Background] Gummerer M, Kummann M, Gratl A, Haller D, Frech A, Klocker J, Fraedrich G, Gruber H. Ultrasound-Guided Fibrin Glue Injection for Treatment of Iatrogenic Femoral Pseudoaneurysms. Vasc Endovascular Surg. 2020 Aug;54(6):497-503. doi: 10.1177/1538574420934631. Epub 2020 Jun 19. PMID 32552570
- [Background] Cope C, Zeit R. Coagulation of aneurysms by direct percutaneous thrombin injection. AJR Am J Roentgenol. 1986 Aug;147(2):383-7. doi: 10.2214/ajr.147.2.383. PMID 3487958
- [Background] Liu W, Liu C, Lu SY. Percutaneous suture technique with ProGlide to manage vascular access pseudoaneurysm after percutaneous coronary intervention procedure: A case report. Chin J Traumatol. 2020 Feb;23(1):34-37. doi: 10.1016/j.cjtee.2019.11.002. Epub 2019 Dec 18. PMID 31956042
- [Background] Kang SS, Labropoulos N, Mansour MA, Baker WH. Percutaneous ultrasound guided thrombin injection: a new method for treating postcatheterization femoral pseudoaneurysms. J Vasc Surg. 1998 Jun;27(6):1032-8. doi: 10.1016/s0741-5214(98)70006-0. PMID 9652465
- [Background] Kurzawski J, Janion-Sadowska A, Zandecki L, Sadowski M. Comparison of the Efficacy and Safety of Two Dosing Protocols for Ultrasound Guided Thrombin Injection in Patients with Iatrogenic Femoral Pseudoaneurysms. Eur J Vasc Endovasc Surg. 2020 Jun;59(6):1019-1025. doi: 10.1016/j.ejvs.2020.01.009. Epub 2020 Feb 1. PMID 32014339